CLINICAL TRIAL: NCT05399004
Title: Sexual Function in Women After Radical Cystectomy
Brief Title: Evaluating Sexual Function in Women Undergoing a Radical Cystectomy for Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen A. Boorjian, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 19-007376; NCI-2021-13603 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-05-26; First posted 2022-06-01 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey): Patients complete surveys over 15-20 minutes at baseline and at 3, 6, and 12 months.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete surveys

SUMMARY:
This study evaluates the general physical, emotional, and sexual function in women undergoing a radical cystectomy for bladder cancer. A radical cystectomy is a surgical procedure that involves the removal of the bladder, uterus, ovaries, fallopian tubes, and part of the vagina. This may affect sexual function in women. This study seeks to understand how radical cystectomy alters sexual function and well-being, and what factors may affect this change.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize pre-operative sexual function and interest in sexual activity of women undergoing radical cystectomy.

II. To identify patient understanding and expectations as they relate to sexual dysfunction after radical cystectomy.

III. To describe pre-operative importance in sexual function recovery after radical cystectomy.

IV. Quantify the changes in sexual function within the year following radical cystectomy in women.

V. Explore the effects of age, baseline sexual function, general quality of life, parity, menopausal status, hormone replacement therapy (topical versus [vs.] oral), general and cancer related quality of life, chemotherapy (neoadjuvant vs. adjuvant), treatment-related complications and performance status on sexual function outcomes.

VI. Explore the effects of robotic vs. open approach, extracorporeal vs. intracorporal approach, organ-sparing (ovaries, uterus, cervix, anterior vaginal wall), type of vaginal closure (vertical vs. horizontal), nerve sparing, urinary diversion type (ileal conduit vs. neobladder vs. continent cutaneous diversion) on sexual function outcomes.

VII. Quantify the changes in sexual activity interest within the year following radical cystectomy.

OUTLINE:

Patients complete surveys over 15-20 minutes at baseline and at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult women greater than 18 years of age
* A diagnosis of bladder cancer
* Planned to undergo a radical cystectomy
* Willing and able to complete survey questionnaires

Exclusion Criteria:

* Inability to provide informed consent
* Non-English speaking
* Life expectancy less than 2 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients undergoing radical cystectomy for bladder cancer between September 1, 2019 and December 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Preoperative sexual function | Baseline
  Assessed using the Patient Reported Outcomes Measurement Information System (PROMIS) Brief Profile Sexual Function and Satisfaction version 2 (v2.0). Will utilize descriptive statistics to report preoperative sexual function. Frequencies and percentages will be reported for categorical variables and mean (standard deviation) or median (interquartile range) for continuous variables.
Interest in sexual activity | From baseline to 3, 6, and 12 months
  Will descriptively summarize the within-patient changes using the PROMIS Brief Profile Sexual Function and Satisfaction v2.0. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Lubrication | From baseline to 3, 6, and 12 months
  Will descriptively summarize the within-patient changes using the PROMIS Brief Profile Sexual Function and Satisfaction v2.0. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Vaginal discomfort | From baseline to 3, 6, and 12 months
  Will descriptively summarize the within-patient changes using the PROMIS Brief Profile Sexual Function and Satisfaction v2.0. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Satisfaction with sex life | From baseline to 3, 6, and 12 months
  Will descriptively summarize the within-patient changes using the PROMIS Brief Profile Sexual Function and Satisfaction v2.0. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.

SECONDARY OUTCOMES:
Labial discomfort | From baseline to 3, 6, and 12 months
  Will descriptively summarize the within-patient changes using the PROMIS Brief Profile Sexual Function and Satisfaction v2.0. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Clitoral discomfort | From baseline to 3, 6, and 12 months
  Will descriptively summarize the within-patient changes using the PROMIS Brief Profile Sexual Function and Satisfaction v2.0. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Orgasm ability | From baseline to 3, 6, and 12 months
  Will descriptively summarize the within-patient changes using the PROMIS Brief Profile Sexual Function and Satisfaction v2.0. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Orgasm pleasure | From baseline to 3, 6, and 12 months
  Will descriptively summarize the within-patient changes using the PROMIS Brief Profile Sexual Function and Satisfaction v2.0. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Change in sexual function scores | From baseline to 12 months
  Will use a linear mixed effects model of 12-month sexual function scores adjusting for baseline function to evaluate independent variables of interest related to the surgical procedure: age, robotic/open approach, pelvic organ sparing and diversion type. Variables of interest will be analyzed separately. In the analysis of robotic vs. open approach, the model will include terms for time (after surgery: 3, 6, and 12 months, using a discrete time formulation), approach (robotic=1, open=0), and approach by time interaction. Contrasts of the interaction and main effects will allow estimation of whether outcomes at 12 months differ by approach.

OTHER OUTCOMES:
Physical function | From baseline to 3, 6, and 12 months
  Assessed using the PROMIS - 29 Profile v2.1. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Fatigue | From baseline to 3, 6, and 12 months
  Assessed using the PROMIS - 29 Profile v2.1. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Pain interference | From baseline to 3, 6, and 12 months
  Assessed using the PROMIS - 29 Profile v2.1. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Depressive symptoms | From baseline to 3, 6, and 12 months
  Assessed using the PROMIS - 29 Profile v2.1. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Anxiety | From baseline to 3, 6, and 12 months
  Assessed using the PROMIS - 29 Profile v2.1. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Ability to participate in social roles and activities | From baseline to 3, 6, and 12 months
  Assessed using the PROMIS - 29 Profile v2.1. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Sleep disturbances | From baseline to 3, 6, and 12 months
  Assessed using the PROMIS - 29 Profile v2.1. Contrasts within the linear mixed effects model will compare changes in subdomain score between different time points.
Preoperative expectations/importance of sexual function recovery | Baseline
  Will use a linear mixed effects model of sexual function scores measured post-baseline through 12 months, adjusted for baseline sexual function score to evaluate if preoperative expectation/importance of sexual function recovery is associated with outcomes over time.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Boorjian, Principal Investigator — Mayo Clinic in Rochester
Locations (14):
- United States (14):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Louisiana State University, Lafayette, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Albany Medical Center, Albany, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Washington Medical Center - Montlake, Seattle, Washington

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials